CLINICAL TRIAL: NCT06023017
Title: The Effect of Preoperative Prone Position Training on Postoperative Pulmonary Complications in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: The Effect of Preoperative Prone Position Training on PPCs in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CQMUAZD2023-2
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pulmonary Complications
Keywords: pulmonary complications, prone position,sleeve gastrectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Position Training group (PPT group) (Experimental): All patients were admitted to our hospital at least 3 days before surgery. Patients in the intervention group (PPT group) received the prone position training daily in the hospital, three times a day, and about 1 hours every times, for at least 3 days before surgery. On the day of admission to the hospital, the patients in the PPT group were instructed to perform prone position training by nurses who were previously trained by prone position training.
  Interventions: Behavioral: Prone Position Training
- Control group (C group) (Placebo Comparator): Patients in the control group (C group) received standard perioperative care without any prone position training.
  Interventions: Behavioral: standard perioperative care without any prone position training

INTERVENTIONS:
Behavioral: Prone Position Training — All patients were admitted to our hospital at least 3 days before surgery. Patients in the intervention group (PPT group) received the prone position training daily in the hospital, three times a day, and about 1 hours every times, for at least 3 days before surgery. On the day of admission to the hospital, the patients in the PPT group were instructed to perform prone position training by nurses who were previously trained by prone position training.
  Arms: Prone Position Training group (PPT group)
Behavioral: standard perioperative care without any prone position training — Patients in the control group (C group) received standard perioperative care without any prone position training.
  Arms: Control group (C group)

SUMMARY:
Postoperative pulmonary complications(PPCs) is a common complication in patients undergoing surgery under general anesthesia, particularly in obese patients. Relevant studies have shown that PPCs are more common in patients undergoing laparoscopic sleeve gastrectomy, which contribute to significant increases in morbidity, mortality, length of postoperative hospital stay and medical consumption. According to some reports, the incidence of PPCs in obese patients after abdominal surgery is about 40%. The reduction in pulmonary volume and respiratory muscular activation after major abdominal surgery due to surgery-related shallow breathing, pain, longterm bed rest, mucociliary clearance disorder, and diaphragmatic dysfunction may be the main causes of PPCs.

Numerous studies have demonstrated physiological improvement related to prone positioning. Prone positioning consists of placing a patient face down. Prone positioning has been used for to improve oxygenation in patients who require invasive mechanical ventilation for acute respiratory distress syndrome (ARDS). It has also been applied to non-intubated patients with acute respiratory failure (ARF), to improve oxygenation and delay or even avoid the need for invasive ventilation. So, the purpose of this study is to observe whether preoperative prone position training can reduce the incidence of pulmonary complications after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Postoperative pulmonary complications(PPCs) is a common complication in patients undergoing surgery under general anesthesia, particularly in obese patients. PPCs refer to the clinical abnormal changes in the lungs after surgery, These include lung infections (pneumonia), atelectasis, pleural effusion, bronchospasm, acute respiratory failure or acute respiratory distress syndrome (ARDS). Postoperative atelectasis could last for more than 24h and contribute to a variety of other complications, including hypoxemia and pneumonia. Relevant studies have shown that PPCs are more common in patients undergoing laparoscopic sleeve gastrectomy, which contribute to significant increases in morbidity, mortality, length of postoperative hospital stay and medical consumption. According to some reports, the incidence of PPCs in obese patients after abdominal surgery is about 40%，and our hospital preliminary investigation, the incidence of PPCs in patients undergoing laparoscopic sleeve gastrectomy is approximately 30%. The reduction in pulmonary volume and respiratory muscular activation after major abdominal surgery due to surgery-related shallow breathing, pain, longterm bed rest, mucociliary clearance disorder, and diaphragmatic dysfunction may be the main causes of PPCs.

Numerous studies have demonstrated physiological improvement related to prone positioning. Prone positioning consists of placing a patient face down. Prone positioning has been used for to improve oxygenation in patients who require invasive mechanical ventilation for acute respiratory distress syndrome (ARDS). It has also been applied to non-intubated patients with acute respiratory failure (ARF), to improve oxygenation and delay or even avoid the need for invasive ventilation.

Currently, the mechanisms of prone position training are decreased lung compression in the gravity dependant zone,homogenisation of transpulmonary pressure, improvement of ventilation/perfusion ratio, and reduction of ventilator-induced lung injury (VILI) or patient self-inflicted lung injury (P-SILI). By placing the patient in the prone position, the lungs compression due to its own weight is reduced via a gravitational-dependent redistribution of fluids. In addition,the weight of the mediastinum is supported by the sternum, the stiffer part of the chest. At the same time, the diaphragm is displaced caudally, decreasing compression of the posterior-caudal lung parenchyma. Finally, in a triangular-shaped lung, more parenchyma is included in the dorsal half than in the ventral one resulting in a more aerated lung in prone positioning.

So, the purpose of this study is to observe whether preoperative prone position training can reduce the incidence of PPCs after laparoscopic sleeve gastrectomy.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement. All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study. This study is a prospective, randomized, controlled clinical trial guided by the standard of good clinical practice (GCP),and eligible participants are divided into two groups: group PPT and group C,and primary assess the incidence of PPCs after laparoscopic sleeve gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Body mass index(BMI)≥30 kg/m2
* Clinical diagnosis of metabolic syndrome, and undergoing Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

* Emergency surgery
* Cognitive dysfunction
* American Society of Anesthesiologists class ≥ IV
* Fractures (face, collarbone, ribs, spine, limbs)
* History of spontaneous pneumothorax
* Increased intracranial pressure
* pregnancy
* Systemic infection
* Patients with hemodynamic instability
* Other conditions that are not suitable for prone position
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications(PPCs) | 3 days after surgery
  The PPCs included pneumonia, atelectasis, pleural effusion, respiratory failure, and unplanned intubations

SECONDARY OUTCOMES:
arterial partial pressure of oxygen (PaO2) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis
arterial partial pressure of carbon dioxide (PaCO2) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis
oxygenation index (OI) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis
extubation time | 1 Day of surgery
  extubation time in postanesthesia care unit(PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China